CLINICAL TRIAL: NCT03126370
Title: Effects of Ledipasvir/Sofosbuvir Treatment on the Pharmacokinetics and Renal Safety of Tenofovir Alafenamide (TAF) in Patients With HIV.
Brief Title: Effects of Ledipasvir/Sofosbuvir on the Pharmacokinetics and Renal Safety of Tenofovir Alafenamide (TAF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-0490
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C; HIV Coinfection
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; emtricitabine tenofovir alafenamide; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAF with a boosted PI and LDV/SOF (Experimental): Participants who are already taking tenofovir disoproxil fumarate 300 mg (in the form of Viread or Truvada) in combination with either a ritonavir- or cobicistat-boosted protease inhibitor for HIV treatment will continue to take their prescribed treatment for 12 weeks after enrollment.
  Participants will be switched from tenofovir disoproxil fumarate to tenofovir alafenamide (TAF) 25 mg/emtricitabine (FTC) 200 mg (Descovy) with a boosted protease inhibitor for the next 12 weeks.
  After taking TAF/FTC for 12 weeks, participants will then start taking ledipasvir 90mg/sofosbuvir 400mg (LDV/SOV, Harvoni) in combination with TAF/FTC and a boosted protease inhibitor for 4 weeks.
  Participants will then return to taking TAF/FTC with a boosted protease inhibitor for the final 12 weeks of the study.
  Interventions: Drug: TDF with a boosted protease inhibitor; Drug: TAF with a boosted protease inhibitor; Drug: TAF with a boosted protease inhibitor and LDV/SOF

INTERVENTIONS:
Drug: TDF with a boosted protease inhibitor — Participants who are already taking tenofovir disoproxil fumarate 300 mg (in the form of Viread or Truvada) in combination with either a ritonavir- or cobicistat-boosted protease inhibitor for HIV treatment will continue to take their prescribed treatment for 12 weeks after enrollment.
  Other: Blood draws for tenofovir PK, renal function assessment
  Other Names: Viread or Truvada with a boosted protease inhibitor
Drug: TAF with a boosted protease inhibitor — Participants will be switched from tenofovir disoproxil fumarate to tenofovir alafenamide 25 mg/emtricitabine 200 mg with a boosted protease inhibitor.
  Other: Blood draws for tenofovir PK, renal function assessment
  Other Names: Descovy with a boosted protease inhibitor
Drug: TAF with a boosted protease inhibitor and LDV/SOF — After taking tenofovir alafenamide/emtricitabine for 12 weeks, participants will then start taking ledipasvir 90 mg/sofosbuvir 400 mg (Harvoni) in combination with the tenofovir alafenamide 25 mg/emtricitabine 200 mg (Descovy) and a boosted protease inhibitor for 4 weeks. Subjects will then return to taking tenofovir alafenamide 25 mg/emtricitabine 200 mg (Descovy) and a boosted protease inhibitor for the final 12 weeks.
  Other: Blood draws for tenofovir PK, renal function assessment
  Other Names: Descovy with a boosted protease inhibitor and Harvoni

SUMMARY:
This study will evaluate the effect of ledipasvir/sofosbuvir (LDV/SOF) treatment on the pharmacokinetics (PK) and renal safety of tenofovir in the form of tenofovir alafenamide (TAF). Subjects living with human immunodeficiency virus (HIV) who are receiving tenofovir-based antiretroviral therapy (in the form of tenofovir disoproxil fumarate [TDF]), and are also taking a ritonavir- or cobicistat-boosted protease inhibitor will be invited to participate.

The study will consist of five visits: a screening visit, three abbreviated 4-hour pharmacokinetic visits, and one end-of-study follow-up visit.

Subjects will also be asked to use a Wisepill device, which will track medication adherence throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-70 years of age
* Have been taking TDF and a ritonavir- or cobicistat-boosted protease inhibitor as part of standard care for treatment of HIV

Exclusion Criteria:

* eGFR < 30 mL/min
* Pregnant or planning pregnancy
* Breastfeeding
* Any medical, social, or mental-health issue(s) that, in the opinion of the investigators, could interfere with study participation or the study outcomes
* Signs or symptoms of decompensated liver disease
* Hepatitis B infection
* Medications that may cause unwanted drug interactions with ledipasvir/sofosbuvir or emtricitabine/tenofovir alafenamide
* Unwillingness or inability to comply with study procedures
* Chronic hepatitis C infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Kiser, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Not Applicable. As per the question above, we do not plan to share IPD

REFERENCES:
- [Background] Sulkowski MS. Hepatitis C virus-human immunodeficiency virus coinfection. Liver Int. 2012 Feb;32 Suppl 1:129-34. doi: 10.1111/j.1478-3231.2011.02719.x. PMID 22212583
- [Background] Genovese D, Boesecke C, Coppola N, Vella S. Virus Variability and Its Impact on HIV and Hepatitis Therapy. Adv Virol. 2012;2012:607527. doi: 10.1155/2012/607527. Epub 2012 Dec 27. No abstract available. PMID 23326266
- [Background] MacBrayne CE, Kiser JJ. Pharmacologic Considerations in the Treatment of Hepatitis C Virus in Persons With HIV. Clin Infect Dis. 2016 Jul 15;63 Suppl 1(Suppl 1):S12-23. doi: 10.1093/cid/ciw220. PMID 27363437
- [Background] Honer Zu Siederdissen C, Maasoumy B, Marra F, Deterding K, Port K, Manns MP, Cornberg M, Back D, Wedemeyer H. Drug-Drug Interactions With Novel All Oral Interferon-Free Antiviral Agents in a Large Real-World Cohort. Clin Infect Dis. 2016 Mar 1;62(5):561-7. doi: 10.1093/cid/civ973. Epub 2015 Nov 26. PMID 26611779
- [Background] Afdhal N, Reddy KR, Nelson DR, Lawitz E, Gordon SC, Schiff E, Nahass R, Ghalib R, Gitlin N, Herring R, Lalezari J, Younes ZH, Pockros PJ, Di Bisceglie AM, Arora S, Subramanian GM, Zhu Y, Dvory-Sobol H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Sulkowski M, Kwo P; ION-2 Investigators. Ledipasvir and sofosbuvir for previously treated HCV genotype 1 infection. N Engl J Med. 2014 Apr 17;370(16):1483-93. doi: 10.1056/NEJMoa1316366. Epub 2014 Apr 11. PMID 24725238
- [Background] Naggie S, Cooper C, Saag M, Workowski K, Ruane P, Towner WJ, Marks K, Luetkemeyer A, Baden RP, Sax PE, Gane E, Santana-Bagur J, Stamm LM, Yang JC, German P, Dvory-Sobol H, Ni L, Pang PS, McHutchison JG, Stedman CA, Morales-Ramirez JO, Brau N, Jayaweera D, Colson AE, Tebas P, Wong DK, Dieterich D, Sulkowski M; ION-4 Investigators. Ledipasvir and Sofosbuvir for HCV in Patients Coinfected with HIV-1. N Engl J Med. 2015 Aug 20;373(8):705-13. doi: 10.1056/NEJMoa1501315. Epub 2015 Jul 21. PMID 26196665
- [Background] German P GK, Pang PS, et al. Drug Interactions Between the anti-HCV Regimen Ledipasvir/Sofosbuvir and Ritonavir-Boosted Protease Inhibitors plus Emtricitabine/Tenofovir DF. CROI 2015; February 23-26, 2015; Seattle WA.
- [Background] MacBrayne CE MK, Fierer DS, et al. Increase Tenofovir Diphosphate in Red Blood Cells, but Not Tenofovir in Plasma, with Sofosbuvir and Ribavirin. 17th International Workshop on Clinical Pharmacology of HIV and Hepatitis Therapy; Washington DC, June 2016 Accepted Abstract (Oral).
- [Background] Hall AM, Hendry BM, Nitsch D, Connolly JO. Tenofovir-associated kidney toxicity in HIV-infected patients: a review of the evidence. Am J Kidney Dis. 2011 May;57(5):773-80. doi: 10.1053/j.ajkd.2011.01.022. Epub 2011 Mar 23. PMID 21435764
- [Background] Tourret J, Deray G, Isnard-Bagnis C. Tenofovir effect on the kidneys of HIV-infected patients: a double-edged sword? J Am Soc Nephrol. 2013 Oct;24(10):1519-27. doi: 10.1681/ASN.2012080857. Epub 2013 Sep 19. PMID 24052632
- [Background] Monteiro N, Branco M, Peres S, Borges F, Mansinho K. The impact of tenofovir disoproxil fumarate on kidney function: four-year data from the HIV-infected outpatient cohort. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19565. doi: 10.7448/IAS.17.4.19565. eCollection 2014. PMID 25394072
- [Background] Moss DM, Neary M, Owen A. The role of drug transporters in the kidney: lessons from tenofovir. Front Pharmacol. 2014 Nov 11;5:248. doi: 10.3389/fphar.2014.00248. eCollection 2014. PMID 25426075
- [Background] Ruane PJ, DeJesus E, Berger D, Markowitz M, Bredeek UF, Callebaut C, Zhong L, Ramanathan S, Rhee MS, Fordyce MW, Yale K. Antiviral activity, safety, and pharmacokinetics/pharmacodynamics of tenofovir alafenamide as 10-day monotherapy in HIV-1-positive adults. J Acquir Immune Defic Syndr. 2013 Aug 1;63(4):449-55. doi: 10.1097/QAI.0b013e3182965d45. PMID 23807155
- [Background] Sax PE, Zolopa A, Brar I, Elion R, Ortiz R, Post F, Wang H, Callebaut C, Martin H, Fordyce MW, McCallister S. Tenofovir alafenamide vs. tenofovir disoproxil fumarate in single tablet regimens for initial HIV-1 therapy: a randomized phase 2 study. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):52-8. doi: 10.1097/QAI.0000000000000225. PMID 24872136
- [Background] Garrison K ea. Drug Interactions between anti-HCV Antivirals Ledipasvir/Sofosbuvir and Integrase Strand Transfer Inhibitor-Based Regimens. 16th International Workshop on Clinical Pharmacology of HIV and Hepatitis Therapy, Washington DC. May 26-28, 2015, abstrac #71
- [Background] Cope R PA, Glowa T, Faulds S, Veldkamp P, Prasad R. Majority of HIV/HCV Co-infected Patients Require Antiretroviral Therapy Switch Prior to Use of Simeprevir (abstract 651). CROI 2015; February 23-26, 2015. Seattle, WA.
- [Background] Langness J LB, Rogers M, J. KJ. Readying HIV/HCV Coinfected Patients for HCV Treatment: Occurrence and Management of Antiviral Interactions (abstract 18). 16th International Workshop on Clinical Pharmacology of HIV and Hepatitis Therapy; May 26-28, 2015; Washington, DC.
- [Background] Havens PL, Kiser JJ, Stephensen CB, Hazra R, Flynn PM, Wilson CM, Rutledge B, Bethel J, Pan CG, Woodhouse LR, Van Loan MD, Liu N, Lujan-Zilbermann J, Baker A, Kapogiannis BG, Gordon CM, Mulligan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 063 Study Team. Association of higher plasma vitamin D binding protein and lower free calcitriol levels with tenofovir disoproxil fumarate use and plasma and intracellular tenofovir pharmacokinetics: cause of a functional vitamin D deficiency? Antimicrob Agents Chemother. 2013 Nov;57(11):5619-28. doi: 10.1128/AAC.01096-13. Epub 2013 Sep 3. PMID 24002093
- [Background] Bushman LR, Kiser JJ, Rower JE, Klein B, Zheng JH, Ray ML, Anderson PL. Determination of nucleoside analog mono-, di-, and tri-phosphates in cellular matrix by solid phase extraction and ultra-sensitive LC-MS/MS detection. J Pharm Biomed Anal. 2011 Sep 10;56(2):390-401. doi: 10.1016/j.jpba.2011.05.039. Epub 2011 Jun 6. PMID 21715120
- [Background] Anderson PL, Kiser JJ, Gardner EM, Rower JE, Meditz A, Grant RM. Pharmacological considerations for tenofovir and emtricitabine to prevent HIV infection. J Antimicrob Chemother. 2011 Feb;66(2):240-50. doi: 10.1093/jac/dkq447. Epub 2010 Nov 30. PMID 21118913
- [Background] Anderson PL, Glidden DV, Liu A, Buchbinder S, Lama JR, Guanira JV, McMahan V, Bushman LR, Casapia M, Montoya-Herrera O, Veloso VG, Mayer KH, Chariyalertsak S, Schechter M, Bekker LG, Kallas EG, Grant RM; iPrEx Study Team. Emtricitabine-tenofovir concentrations and pre-exposure prophylaxis efficacy in men who have sex with men. Sci Transl Med. 2012 Sep 12;4(151):151ra125. doi: 10.1126/scitranslmed.3004006. PMID 22972843
- [Background] Anderson PL, Glidden DV, Bushman LR, Heneine W, Garcia-Lerma JG. Tenofovir diphosphate concentrations and prophylactic effect in a macaque model of rectal simian HIV transmission. J Antimicrob Chemother. 2014 Sep;69(9):2470-6. doi: 10.1093/jac/dku162. Epub 2014 May 26. PMID 24862094
- [Background] Kiser JJ, Fletcher CV, Flynn PM, Cunningham CK, Wilson CM, Kapogiannis BG, Major-Wilson H, Viani RM, Liu NX, Muenz LR, Harris DR, Havens PL; Adolescent Trials Network for HIV/AIDS Interventions. Pharmacokinetics of antiretroviral regimens containing tenofovir disoproxil fumarate and atazanavir-ritonavir in adolescents and young adults with human immunodeficiency virus infection. Antimicrob Agents Chemother. 2008 Feb;52(2):631-7. doi: 10.1128/AAC.00761-07. Epub 2007 Nov 19. PMID 18025112
- [Background] Kiser JJ, Aquilante CL, Anderson PL, King TM, Carten ML, Fletcher CV. Clinical and genetic determinants of intracellular tenofovir diphosphate concentrations in HIV-infected patients. J Acquir Immune Defic Syndr. 2008 Mar 1;47(3):298-303. doi: 10.1097/qai.0b013e31815e7478. PMID 18398970
- [Background] Kiser JJ, Carten ML, Aquilante CL, Anderson PL, Wolfe P, King TM, Delahunty T, Bushman LR, Fletcher CV. The effect of lopinavir/ritonavir on the renal clearance of tenofovir in HIV-infected patients. Clin Pharmacol Ther. 2008 Feb;83(2):265-72. doi: 10.1038/sj.clpt.6100269. Epub 2007 Jun 27. PMID 17597712
- [Background] Castillo-Mancilla J, Coyle R, Zheng J, al e. Tenofovir Diphosphate Arising from TAF is Quantifiable in Dried Blood Spots. Conference on Retroviruses and Opportunistic Infections. Seattle Washington, February 13-16, 2017.

RESULTS

PARTICIPANT FLOW:
Groups:
- TAF With a Boosted PI and LDV/SOF: Subjects who are already taking tenofovir disoproxil fumarate 300 mg (in the form of Viread or Truvada) in combination with either a ritonavir- or cobicistat-boosted protease inhibitor for HIV treatment will continue to take their prescribed treatment for 12 weeks after enrollment.
  Subjects will be switched from tenofovir disoproxil fumarate to tenofovir alafenamide (TAF) 25 mg/emtricitabine (FTC) 200 mg (Descovy) with a boosted protease inhibitor for the next 12 weeks.
  After taking TAF/FTC for 12 weeks, subjects will then start taking ledipasvir 90mg/sofosbuvir 400mg (Harvoni) in combination with TAF/FTC and a boosted protease inhibitor for 4 weeks.
  Subjects will then return to taking TAF/FTC with a boosted protease inhibitor for the final 12 weeks of the study.
  TDF with a boosted protease inhibitor: Subjects who are already taking tenofovir disoproxil fumarate 300 mg (in the form of Viread or Truvada) in combination with either a ritonavir- or cobicistat-boosted protease
Period: TDF With a Boosted PI
Arm/Group | TAF With a Boosted PI and LDV/SOF
Started | 10
Completed | 10
Not Completed | 0
Period: TAF With a Boosted PI
Arm/Group | TAF With a Boosted PI and LDV/SOF
Started | 10
Completed | 10
Not Completed | 0
Period: TAF With a Boosted PI and LDV/SOF
Arm/Group | TAF With a Boosted PI and LDV/SOF
Started | 10
Completed | 10
Not Completed | 0
Period: TAF With a Boosted PI
Arm/Group | TAF With a Boosted PI and LDV/SOF
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TAF With a Boosted PI and LDV/SOF
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
eGFR [Mean (Standard Deviation); unit: mL/min/1.73^m2] | 91.5 (26.6)
Weight [Mean (Standard Deviation); unit: kg] | 88.8 (16.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 12 Plasma Tenofovir Area Under the Plasma Concentration vs. Time Curve From Time 0 to 24 Hours (AUC0-24) at 24 and 28 Weeks
Description: Compare plasma tenofovir AUC0-24 between TAF with boosted PI vs. TDF with boosted PI (Phase 2 vs. 1), and between TAF with boosted PI and LDV/SOF vs. TDF with boosted PI (Phase 3 vs. 1)
Time Frame: 12 weeks and 24 weeks and 28 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- TDF With a Boosted PI: Tenofovir disoproxil fumarate with a boosted protease inhibitor
- TAF With a Boosted PI: Tenofovir alafenamide with a boosted protease inhibitor
- TAF With a Boosted PI and LDV/SOF: Tenofovir alafenamide with a boosted protease inhibitor and ledipasvir/sofosbuvir
Arm/Group | TDF With a Boosted PI | TAF With a Boosted PI | TAF With a Boosted PI and LDV/SOF
Number analyzed (Participants) | 10 | 10 | 10
ng*h/mL | 3466 (51.4) | 743 (35.8) | 868 (40.8)

2. Primary Outcome: Change From Week 12 Tenofovir-diphosphate (TFV-DP) in Peripheral Blood Mononuclear Cells (PBMCs) at 24 and 28 Weeks
Description: Compare tenofovir-diphosphate (TFV-DP) in peripheral blood mononuclear cells (PBMCs) between TAF with a boosted PI vs. TDF with a boosted PI (Phase 2 vs. 1), and TAF with a boosted PI and LDV/SOF vs. TDF with a boosted PI (Phase 3 vs. 1).
Time Frame: 12 weeks, and 24 weeks and 28 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fmol/10^6 cells
Arm/Group | TDF With a Boosted PI | TAF With a Boosted PI | TAF With a Boosted PI and LDV/SOF
Number analyzed (Participants) | 10 | 10 | 10
fmol/10^6 cells | 83.0 (66.6) | 926 (23.4) | 1129 (34.9)

3. Secondary Outcome: Change From Week 12 Tenofovir-diphosphate (TFV-DP) in Dried Blood Spots (DBS)
Description: Compare tenofovir diphosphate (TFV-DP) in dried blood spots (DBS) between TAF with a boosted PI vs. TDF with a boosted PI (Phase 2 vs. 1), and TAF with a boosted PI and LDV/SOF vs. TDF with a boosted PI (Phase 3 vs. 1)
Time Frame: 12 weeks and 24 and 28 weeks
Population: Comparisons between study phases were controlled for 3-month adherence. Results reported
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fmol/2x7mm punches
Arm/Group | TDF With a Boosted PI | TAF With a Boosted PI | TAF With a Boosted PI and LDV/SOF
Number analyzed (Participants) | 10 | 10 | 10
fmol/2x7mm punches | 36014 (46.4) | 6735 (45.0) | 6100 (41.0)

4. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) and Renal Biomarkers: eGFR
Description: Change in estimated glomerular filtration rate (eGFR)
Time Frame: 12 weeks, 24 weeks, and 28 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min/1.73 m^2
Arm/Group | TDF With a Boosted PI | TAF With a Boosted PI | TAF With a Boosted PI and LDV/SOF
Number analyzed (Participants) | 10 | 10 | 10
mL/min/1.73 m^2 | 86.7 (27.6) | 91.0 (23.0) | 88.1 (24.9)

5. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) and Renal Biomarkers: UPCR
Description: Change in estimated glomerular filtration rate (eGFR) and renal biomarkers: Urine protein to creatinine ratio (UPCR)
Time Frame: 12 weeks, 24 weeks, and 28 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/g
Arm/Group | TDF With a Boosted PI | TAF With a Boosted PI | TAF With a Boosted PI and LDV/SOF
Number analyzed (Participants) | 10 | 10 | 10
mg/g | 134 (65.7) | 118 (50.2) | 97.3 (41.0)

6. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) and Renal Biomarkers: B2M/Cr Ratio, and RBP/Cr Ratio
Description: Change in renal biomarkers: urinary beta-2 microglobulin (B2M)/creatinine (Cr) ratio, and urinary retinol binding protein (RBP)/Cr ratio
Time Frame: 12 weeks, 24 weeks, and 28 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/g
Arm/Group | TDF With a Boosted PI | TAF With a Boosted PI | TAF With a Boosted PI and LDV/SOF
Number analyzed (Participants) | 10 | 10 | 10
ug/g
  β2M:Cr ratio | 419 (176) | 224 (167) | 178 (156)
  RBP:Cr ratio | 436 (174) | 242 (180) | 146 (91.6)

ADVERSE EVENTS:
Time Frame: 40 weeks
Description: Adverse events were graded according to the Division of AIDS AE Reporting Table (July 2017, version 2.1)
Arm/Group | TDF With a Boosted PI | TAF With a Boosted PI | TAF With a Boosted PI and LDV/SOF
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF With a Boosted PI (N=10) | TAF With a Boosted PI (N=10) | TAF With a Boosted PI and LDV/SOF (N=10)
Renal events deemed possibly, probably or related (Renal and urinary disorders) | 2 (3) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT03126370/Prot_SAP_000.pdf